CLINICAL TRIAL: NCT00004886
Title: Phase I Study to Determine the Safety of MS-209 in Combination With Docetaxel in Patients With a Solid Progressive Tumor
Brief Title: MS 209 Plus Docetaxel in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16992; EORTC-16992
Record Dates: First submitted 2000-03-07; First posted 2003-10-01 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Docetaxel

INTERVENTIONS:
Drug: docetaxel
Drug: dofequidar fumarate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of MS 209 plus docetaxel in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of oral MS-209 when given with docetaxel IV in patients with advanced solid malignant tumors.
* Assess the toxicity of this regimen in these patients.

OUTLINE: This is a dose escalation, multicenter study of MS-209.

Patients receive docetaxel IV over 1 hour on day 1 of a 3 week course. On day 1 of the 2nd course, patients receive MS-209 orally followed by docetaxel IV over 1 hour. Treatment is repeated every 3 weeks for 4-7 courses (including course with docetaxel alone). Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of MS-209 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 3 or 3 of 6 patients experience dose limiting toxicities.

Patients are followed every 6 weeks.

PROJECTED ACCRUAL: Approximately 3-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced malignant solid tumor

  * No gastric cancer
* No brain involvement or leptomeningeal disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 11.2 g/dL

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.4 mg/dL

Cardiovascular:

* Normal cardiac function
* Left ventricular ejection fraction normal

Other:

* No digestive disease that hampers absorption
* No unstable systemic disease or uncontrolled infection that precludes study
* No psychological, familial, sociological, or geographical condition that precludes compliance
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No prior docetaxel
* No other concurrent chemotherapy

Endocrine therapy:

* At least 4 weeks since prior hormonal therapy

Radiotherapy:

* At least 4 weeks since prior radiotherapy (6 weeks if extensive)

Surgery:

* Not specified

Other:

* No other concurrent anticancer drugs
* No other concurrent investigational therapies
* No H2-blockers, proton pump inhibitors, sucralfate or any other drug that would impair absorption
* No concurrent drugs exhibiting liver, kidney, heart or lung toxicity
* No concurrent MDR-modulating drugs (e.g., calcium antagonists, immunosuppressives)
* No concurrent antifungals (ketoconazole, fluconazole) or antibiotics (clarithromycin, erthromycin) that interfere with MS-209 metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1999-12; Primary Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Dieras, MD, Study Chair — Institut Curie
Locations (3):
- France (2):
  - Centre Oscar Lambret, Lille
  - Institut Curie - Section Medicale, Paris
- Haemato-Onkologische Praxis und Tagesklinik, Munich (Muenchen), Germany